CLINICAL TRIAL: NCT06865014
Title: Changes in Sleep Patterns, Dietary Intake, Cognitive Skills, Anticipation Time and Physical Activity Levels During Ramadan in Healthy Young Women
Brief Title: Cognitive and Psychomotor Skills and Behavioural Changes During Ramadan in Women
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ümid Karlı, Professor, Abant Izzet Baysal University
Other Study IDs: BAIBU-SBF-UK-02
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Fasting, Intermittent; Food Habits; Sleep
Keywords: Physical Fitness; Body Composition; Cognitive Skills; Ramadan Fasting; Anticipation Time
MeSH Terms: conditions — Intermittent Fasting; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ramadan Intermittent Fasting Group: Twenty two healthy, moderately active young women who regularly fast during Ramadan.
  Interventions: Other: Intermittent Ramadan Fasting

INTERVENTIONS:
Other: Intermittent Ramadan Fasting — Intermittent fasting during the month Ramadan

SUMMARY:
This study will observe the participants fasting during the month ramadan. Descriptive characteristics and assessments of sleep, food consumption, body composition, cognitive skills, anticipation time, and physical activity will be conducted before, during and after ramadan.

DETAILED DESCRIPTION:
The aim of this is investigating the changes in sleep patterns, dietary intake, cognitive skills, anticipation time and physical activity levels during Ramadan in healthy young women.

After giving information about the research, participants' descriptive characteristics such as age, height, body weight, body fat percentage, and chronotype (Morningness-Eveningness Questionnaire) will be determined and recorded. Participants' sleep patterns (Actigraphy and Pittsburgh Sleep Quality Index), food consumption (BEBIS), cognitive skills (Stroop test, Letter digit test), anticipation time (Bassin Anticipation Timer), and physical activity levels (International Physical Activity Questionnaire) will be assessed before Ramadan (Pre-R), in the first week of Ramadan (FW-R), in the last week of Ramadan (LW-R) and after Ramadan (Post-R). Additionally, body composition measurements will be taken in Pre-R, LW-R and Post-R. The completion of questionnaires and scales will be conducted individually in a quiet environment. Sleep records will be obtained using an actigraphy device in the participants' own sleep environments. Other measurements will be conducted at the University Performance and Exercise Physiology Laboratory under controlled temperature (22-24°C) and humidity (50-60%).

ELIGIBILITY:
Inclusion Criteria:

* Voluntariness: Participants must be willing to participate in the study voluntarily and provide informed consent.
* Absence of any health issues
* No chronic sleep problems
* No use of sleep medication
* Fasting throughout the study period during the month Ramadan

Exclusion Criteria:

* Complications During the Intervention: Participants who experience any complications during the month Ramadan while fasting.
* Irregular fasting behavior during Ramadan

Ages: 18 Years to 24 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — This study will focus on female participants.
Study Population: Twenty two healthy, moderately active young women who regularly fast during the month Ramadan will be the participants in this study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2025-02-23 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Actigraphy | Pre-test, following one week first mid-test, following three weeks second mid-test and following two weeks post-test
  Actigraphy is a less invasive method compared to other sleep measurement methods such as polysomnography
Body weight measurement | Pre-test, following one month mid-test and following another one month post-test
  Test that involves measuring body weight using medical scales
Body fat percentage | Pre-test, following one month mid-test and following another one month post-test
  Includes determination of body fat percentage using a bioelectrical impedance analyzer
Food consumption assessment | Pre-test, following one week first mid-test, following three weeks second mid-test and following two weeks post-test
  Participants will be asked to record their food and liquid intake in detail for three consecutive days (two weekdays and one weekend day). All data will then be entered into the nutrition data system, and total energy intake, carbohydrate amount (CHO), protein, fat, and liquid consumption will be calculated.
Stroop test | Pre-test, following one week first mid-test, following three weeks second mid-test and following two weeks post-test
  The Stroop test reflects mainly the frontal lobe activity. The Stroop effect demonstrates an individual's ability to shift perceptual setup according to changing demands, suppress habitual response patterns, and perform unconventional actions, which are primarily related to frontal lobe activity. The test also measures information processing speed.
Letter Digit Substitution Test | Pre-test, following one week first mid-test, following three weeks second mid-test and following two weeks post-test
  The Letter Digit Substitution Test is an adapted matching test developed to measure information processing speed. The test contains a key containing nine letters of the alphabet and the numbers 1 to 9. Then there are randomly arranged letters and participants will be asked to match the random letters with the appropriate number indicated by the key.
Anticipation time measurement | Pre-test, following one week first mid-test, following three weeks second mid-test and following two weeks post-test
  The anticipation time will be measured using the 50575 model of the Bassin Anticipation Timer. The sensitivity of the device will be set to 0.001 seconds, with the anticipation device's speed set to 11 mph (4.9 m/s) and the delay time set to 0-2 seconds. Each participant will undergo 20 measurements per session. Measurements will be manually recorded on the anticipation time measurement sheet.
  The test position for all participants will be standing vertically in front of the anticipation device, with the motion light approaching them. The participant will stand at the end of the device, using their dominant hand to press the stop button at sternum height with one hand. The researcher will hide the start command button behind them to ensure participants cannot see when the test begins. After each trial is recorded, the next trial will be conducted. The fixed anticipation time error (SzSh) and absolute anticipation time error (SzMh) will be automatically calculated.
Physical activity level assessment | Pre-test, following one week first mid-test, following three weeks second mid-test and following two weeks post-test
  The International Physical Activity Questionnaire (IPAQ) will be used to determine their level of physical activity levels. The questionnaire consists of sections that inquire about vigorous physical activity, moderate physical activity, and walking activities of at least 10 minutes duration over the past seven days.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Pre-test, following one month mid-test and following another one month post-test
  Pittsburgh Sleep Quality Index assesses various sleep-related factors, including sleep latency, sleep duration, sleep efficiency, and daytime sleepiness. It is a 19-item self-report questionnaire. Each item is scored from 0 to 3, and the total score ranges from 0 to 57. Higher scores indicate poorer sleep quality.
Chronotype assessment | Only once in the pre-test
  Morningness-Eveningness Questionnaire (MEQ) will be used to assess Chronotype. The form consists of 19 questions, each offering four possible answers. Participants receive different scores based on their responses: questions 3, 4, 5, 6, 7, 8, 9, 13, 14, 15, and 16 are scored between 1 and 4, questions 1, 2, 10, 17, and 18 are scored between 1 and 5, questions 11 and 19 are scored between 0 and 6, and question 12 is scored between 0 and 5. The scores range from 16 to 86, with lower scores indicating evening types and higher scores indicating morning types. Based on the total score, individuals are classified as evening types (16-41 points), intermediate types (42-58 points), and morning types (59-86 points).

CONTACTS AND LOCATIONS:
Overall Officials: Umid Karli, PhD, Principal Investigator — Bolu Abant İzzet Baysal University, Faculty of Sport Sciences, Department of Coaching Education
Locations (1):
- Bolu Abant İzzet Baysal University, Faculty of Sport Sciences,, Bolu, Turkey (Türkiye)